CLINICAL TRIAL: NCT00165373
Title: A Phase I, Safety, Pharmacokinetic and Pharmacodynamic Study of rhEndostatin Protein Administered by Continuous Intravenous Infusion to Pediatric Patients With Cancer
Brief Title: rhEndostatin Protein Involving Pediatric Patients With Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of drug supply
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Mark Kieran, MD, PhD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-222
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Solid Tumors
Keywords: pediatric solid tumors; rhEndostatin
MeSH Terms: interventions — Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rhEndostatin — Given by continuous infustion for 28 days (one of two dosing groups) for a total of 2 cycles. Treatment can be extended if tolerated well.

SUMMARY:
The purpose of this study is to assess the safety of rhEndostatin, to determine how much of the drug stays in the patients blood (pharmacokinetics), to assess the development of proteins in the blood that are produced by the body (antibodies)using rhEndostatin, to determine the effect of rhEndostatin on the formation of new blood vessel factors, and to perform an analysis of the effect of rhEndostatin on circulating endothelial precursor cells (cells in the body that help the tumor build more blood vessels).

DETAILED DESCRIPTION:
* Patients will receive rhEndostatin intravenously continuously for 28 days and will be enrolled into one of 2 dosing groups.
* During the initial course of treatment, subjects will be evaluated for treatment-related side effects. If there are no side effects or disease progression, they may receive an additional 28 days of continuous rhEndostatin.
* During the infusion of rhEndostatin, blood samples will be collected before, during and after the drug is given to determine how much of the drug stays in the blood. Blood will be drawn on days 1, 8, 22 and 29. After the completion of therapy, a blood sample will be collected at least 3 days after to determine the level (if any) of rhEndostatin still in the patients blood.
* Blood and/or urine samples to determine immune reactions against rhEndostatin as well as molecules that tumors may use to stimulate new blood vessel growth will be drawn at the start of the study as well as after the completion of each 28-day cycle and completion of the study.
* When a tumor-specific marker that can be used to monitor the status of the disease is present, blood samples for the measurement marker will be obtained at the start of the study as well as after each cycle.
* Appropriate imaging studies (MRI, CT scan, x-ray) will be done after the completion of the first two 28-day cycles and then at the completion of each 28-day cycle for the duration of therapy.
* Treatment will be continued for 1 year and may be extended if the drugs are well tolerated and disease progression has not occured.

ELIGIBILITY:
Inclusion Criteria:

* Must have had a histological verification of solid tumor at the original diagnosis. For patients with brain stem gliomas and optic pathway tumors, the requirement for histological evaluation may be waived. The patient's disease must be considered refractory to conventional/standard therapy, or a disease for which no conventional therapy exists and is progressive. Patients must have measurable disease for this study.
* Agree to having a central venous access placed
* Be between 2 and 18, inclusive, years of age
* Aspartate aminotransferase and alanine aminotransferase less than 2.5 x ULN-
* Total bilirubin less than 2.0 x ULN
* Serum creatinine less than 2.0 mg/dL or a creatinine clearance or glomerular filtration rate less than 2 times normal for age
* Absolute neutrophil count greater than or equal to 1,000/mm3
* Platelets greater than or equal to 100,000/mm3 (transfusion independent)
* Hemoglobin greater than 8.0 g/dL
* Have an estimated life expectancy of at least 3 months
* Have a Karnofsky performance status greater than 50 for patients aged 10 years or older and a Lansky performance status greater than 50 for patients aged 2 to less than 10 years
* Patients are required to have had an EKG, echocardiogram, and pulse oximetry within age-appropriate levels prior to starting therapy.
* If a woman or man of child producing potential, agree to use effective contraceptive methods (A negative pregnancy test within 72 hours before the administration of rhEndostatin protein will be required for women of childbearing potential.)

Exclusion Criteria:

* Patients with leukemia
* Be pregnant or nursing
* Have a history of bleeding diathesis, hypercoagulable condition, or an active bleeding disorder
* Have any condition that is likely to interfere with regular follow-up
* Have participated in any clinical trial involving conventional or investigational drugs or devices within 4 weeks prior to rhEndostatin protein administration
* Have received radiotherapy or chemotherapy within 4 weeks prior to rhEndostatin protein administration
* Have received nitrosourea or mitomycin C less than 6 weeks prior to initiation of therapy
* Be receiving concurrent treatment with therapeutic doses of heparin or enoxaparin sodium (Lovenox®) (rhEndostatin protein has a heparin binding domain.)
* Have had major surgery within 2 weeks of starting rhEndostatin protein administration This does not include placement of a vascular access device.
* Have a history of bone marrow transplantation or extensive radiotherapy (craniospinal, total body, or radiotherapy to more than half of the pelvis) within the previous 4 months
* Have ionized calcium levels below the lower limits of normal
* Have a history of myocardial infarction within the last 6 months, angina pectoris/angina equivalent in the last 6 months (the patient may be on antianginal medications if the symptoms can be entirely controlled), or have uncontrolled congestive heart failure
* Have an active infection
* Have additional uncontrolled serious medical or psychiatric illness

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety of rhEndostatin protein in pediatric patients with recurrent or progressive cancer that is measurable and that is refractory to standard therapies. | 3 years

SECONDARY OUTCOMES:
To determine how much of the drug stays in the blood of patients (pharmacokinetics)and to evaluate tumor response after treatment with rhEndostatin on this patient population. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Kieran, MD,PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States